CLINICAL TRIAL: NCT02079688
Title: A Phase IIa, Single-centre, Randomised, Vehicle Controlled, Double-blind Trial for Assessment of Efficacy, Safety and Tolerability of the Topical Formulation SB011 Containing a Human GATA-3 Specific DNAzyme and of Systemic Absorption of hgd40 Following Application to Lesional Skin in Patients With Atopic Eczema
Brief Title: Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of the Topical Formulation SB011 Applied to Lesional Skin in Patients With Atopic Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sterna Biologicals GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB011/02/2013
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Mild to Moderate Atopic Dermatitis
Keywords: Antisense oligonucleotide; atopic eczema; atopic dermatitis; Phase II; Transcription factor GATA-3; dermal application; Proof-of-Concept
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SB011, 2 % (Water/Oil/Water) emulsion of hgd40 (Experimental): All patients will perform treatment with formulation SB011 containing 2 % hgd40 and the active ingredient-free vehicle. The comparison of the IMPs will be performed intraindividually.
  Comparison and random assignment of treatments to two distinct treatment areas (area 1, area 2).
  IMP SB011: Topical application of approximately 5 mg/cm2 (250 μl) per treatment area (50 cm2) twice daily on 14 consecutive days, one single last application at the site on Day 15 (29 treatments) daily dosage: Approximately 10 mg hgd40 total dosage: Approximately 145 mg hgd40
  Interventions: Drug: SB011, 2 % (Water/Oil/Water) emulsion of hgd40
- Multiple W/O/W formulation, active ingredient-free vehicle (Placebo Comparator): All patients will perform treatment with formulation SB011 containing 2 % hgd40 and the active ingredient-free vehicle. The comparison of the IMPs will be performed intraindividually.
  Comparison and random assignment of treatments to two distinct treatment areas (Area 1, Area 2).
  Vehicle: Topical application of approximately 5 mg/cm2 (250 μl) per treatment area (50 cm2) twice daily on 14 consecutive days, one single last application at the site on Day 15 (29 treatments)
  Interventions: Drug: Multiple W/O/W formulation, active ingredient-free vehicle

INTERVENTIONS:
Drug: SB011, 2 % (Water/Oil/Water) emulsion of hgd40 — Treatment will be performed BID on 14 consecutive days and one single last application at the site on Day 15 (29 applications in total).
  Two preferably disseminated and contralateral, comparable lesional treatment areas of approximately 50 cm2 each and located on arms, legs, chest, stomach or neck will be chosen. All patients will perform treatment with both formulation SB011 containing 2% hgd40 and the active ingredient-free vehicle. Comparison of the IMPs will be performed intraindividually.
  Approximately 5 mg/cm2 (250 μl) of SB011 (2% hgd40) and the vehicle will be applied to the respective treatment areas. The time between the two applications should include min. 8 hours and max. 16 hours. Patients compliance will be controlled by weighing of the IMPs at each visit. On day 1 the application of the IMPs will be demonstrated to the patients at the clinical site. The first treatment as well as the morning treatment on Days 3, 5, 8, 12, and 15 will be carried out at the clinical site
  Other Names: Active drug substance is hgd40
  Arms: SB011, 2 % (Water/Oil/Water) emulsion of hgd40
Drug: Multiple W/O/W formulation, active ingredient-free vehicle — Treatment will be performed BID on 14 consecutive days and one single last application at the site on Day 15 (29 applications in total).
  Two preferably disseminated and contralateral, comparable lesional treatment areas of approximately 50 cm2 each and located on arms, legs, chest, stomach or neck will be chosen. All patients will perform treatment with both formulation SB011 containing 2% hgd40 and the active ingredient-free vehicle. Comparison of the IMPs will be performed intraindividually.
  Approximately 5 mg/cm2 (250 μl) of SB011 (2% hgd40) and the vehicle will be applied to the respective treatment areas. The time between the two applications should include min. 8 hours and max. 16 hours. Patients compliance will be controlled by weighing of the IMPs at each visit. On day 1 the application of the IMPs will be demonstrated to the patients at the clinical site. The first treatment as well as the morning treatment on Days 3, 5, 8, 12, and 15 will be carried out at the clinical site
  Arms: Multiple W/O/W formulation, active ingredient-free vehicle

SUMMARY:
Atopic dermatitis (AD) is a chronic or chronic recurring inflammatory skin disorder. Patients suffer from eczema and often severe pruritus on the affected skin, as well as from frequent complications and secondary infections. Next to a genetically predetermined defect in epidermal barrier function and vegetative dysfunction, AD arises from an upregulation of Th2-modified immune responses inducing increased IgE-antibody production, cytokine secretion and subsequently, local inflammation.

Although standard therapies of AD, modern topical corticosteroids, show a better ratio of therapeutic effects to side effects, they retain a moderate acceptance due to their non-specific action, strict compliance requirements and possible adverse effects. As a newer alternative, calcineurin inhibitors show fewer side effects but raise concerns regarding long term risks including the possibility of skin carcinogenicity. Therefore, medical need remains for novel therapies for this major public health problem, directed in particular at specific early disease-causing mechanisms and/or molecular targets, with an improved efficacy, safety and compliance.

Novel therapeutic strategies for the treatment of chronic inflammatory diseases by targeting early disease-causing mechanisms are a promising approach for the treatment of AD.

The transcription factor GATA-3 represents the key regulatory factor of Th2-driven immune responses. It is indispensable for the differentiation and activation of Th2 cells; it integrates Th2 signals and induces Th2 cytokine expression. The investigational product SB011 contains the DNAzyme hgd40 that targets GATA-3. By cleaving GATA-3 mRNA hgd40 reduces specific cytokine production and thereby reduces key features of allergic airway inflammation.

DNAzymes are completely generated by chemical synthesis and can be produced under Good Manufacturing Practice (GMP) controlled conditions. The DNAzymes are not biological drugs, i.e. they are not generated by use of any living organism including cell culture or bacteria. The molecules are highly water-soluble and will be applied as a water/oil/water (W/O/W) formulation since multiple emulsions have been shown to protect the active ingredient from degradation on the skin and have penetration enhancing properties in comparison to other carrier systems.

This proof-of-concept study will evaluate the efficacy, safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of the topical formulation SB011 containing 2 % hgd40 twice daily (BID) in patients with mild to moderate atopic eczema.

ELIGIBILITY:
Inclusion Criteria:

* Patient oral and written informed consent
* Adult Caucasian patients (male and female) aged 18-69 years (both included);
* Patients smoking ≤ 10 cigarettes/day
* Patient has confirmed diagnosis of atopic dermatitis using the diagnostic features as described by Hanifin and Rajka, initial diagnosis made at least 12 weeks before first treatment;
* SCORAD (12) between 20 and 50 (mild to moderate atopic dermatitis);
* Two comparable lesional areas of approximately 50 cm2 each (difference in modified local SCORAD not greater than 2) on the arms, legs, chest, stomach or neck (distance between the lesions at least 5 cm), clinical condition of atopic eczema mild to moderate defined by a modified local SCORAD between 7 and 10 with 2 parameters scored at least 2 one being the erythema score;
* Patient has to have an increased total IgE;
* Patient has to have an increased specific IgE of at least 1 of the sx1 allergens with CAP classification II [>0.7 KU/l];
* Erythema score from modified local SCORAD for both lesional areas of at least 2;
* TEWL in the lesional areas at least 12 g/m²h, TEWL value differences ≤ 30 % are allowed between both lesional areas (related to the higher TEWL value);
* Except for atopic diseases or asthma like atopic dermatitis or allergic rhinitis assessed as healthy based on a screening examination including medical history, physical examination of the skin, vital signs, and clinical laboratory results;
* The male patient must agree:
* to use two methods of contraception in combination with his female partner, if she is of childbearing potential (At least one of the contraception methods must be a barrier contraception method)
* The female patient must agree:
* to use two methods of contraception in combination with her male partner, if she is of childbearing potential;

Exclusion Criteria:

* History of allergic reactions to any active or inactive component of the IMP;
* Presence of clinically significant diseases other than asthma or atopic diseases (cardiovascular, renal, hepatic, gastrointestinal, haematological, neurological, genitourinary, autoimmune, endocrine, metabolic, etc.) which in the opinion of the investigator, influence the results of the trial or the patient's ability to take part in it;
* Inherent or acquired immune deficiency, immune deficiency in consequence of drug use;
* Immune mediated diseases;
* Suntan, hyperpigmentation or tattoos in the test fields;
* Dark-skinned persons whose skin colour prevents ready assessment of skin reactions;
* Systemic bacterial or mycotic as well as severe viral systemic infections;
* Severe systemic other disease;
* Patients with a resting heart rate <50 and >100 bpm, systolic blood pressure <100 and >150 mmHg, diastolic blood pressure <60 and >95 mmHg;
* UV-therapy within 6 weeks before first treatment and during the trial;
* History or current evidence of a malignant tumour (an excised basal cell carcinoma distant from target lesion with at least 14 days after surgery will be allowed);
* Clinically relevant abnormalities in serology, clinical chemical, haematological or in any other laboratory variables;
* Chronic or acute infections (a small lesion of non-treated onychomycosis will be allowed in the opinion of the investigator);
* Pregnancy or nursing
* Signs of secondary infections on the lesions to be treated;
* History of previous administration of SB011 or any other registered or investigational oligonucleotide-based drug;
* History or presence of alcohol or drug abuse;
* Consumption of alcohol within 48 h before administration of IMPs and during the trial;
* Use of any medication (including over-the-counter medication such as herbal products) except allowed concomitant medication within 2 weeks (for biologics: 6 months, for systemic treatment of atopic dermatitis 4 weeks) before administration of the IMPs or within <10 times the elimination half-life of the respective drug, or the duration of the pharmacodynamics effect, whatever is longer, or anticipated concomitant medication during the treatment period (exception: asthma may be found in patients with AD, therefore the continuation of inhalative treatment with corticosteroids in patients with asthma accompanying AD that began at least four weeks prior to randomisation will be allowed; dose limited: ≤ 300 μg/d fluticasone propionate or equivalent);
* Treatment with known cytochrome P450 enzyme inducing or inhibiting agents (St. John's Wort ("Johanniskraut"), barbiturates, phenothiazines, cimetidine, ketoconazole) within 30 days before administration of the IMPs or during the trial;
* Consumption of grapefruit, grapefruit juice within 14 days prior to the IMP administration or during the trial;
* Need for additional skin care products in the treatment area(s);
* Use of skin care products with anti-septic components during the last four weeks before first treatment and during the trial or anti-septic textiles with contact to the target lesions;
* Proneness to orthostatic dysregulation, faintings, or blackouts;
* Planned donation of germ cells, blood, organs, bone marrow during the course of the trial or within 6 months thereafter;
* Participation in another clinical trial with an investigational drug or device within the last 3 months. For biologics, the minimum exclusion period is at least 6 months or the time of duration of the pharmacodynamics effect or 10 times the half-life of the respective drug whatever is longer before inclusion in this trial;
* Lack of ability or willingness to give informed consent;
* Anticipated non-availability for trial visits/procedures;
* Anticipated lack of willingness or inability to cooperate adequately;
* Close affiliation with the investigators (e.g. a close relative) or with persons working at bioskin GmbH or with persons working at the study site or with employees of sterna biologicals GmbH & Co. KG;
* Vulnerable patients (e.g., persons kept in detention)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change of local SCORing atopic dermatitis (SCORAD) from baseline to Day 15. | On baseline (day 1) and on day 15 (Last day after 2 Weeks IMP administration)
  The following parameters are included in scoring:
  A: the extent of the involved body area;
  B: the intensity of the criteria erythema, edema/papulation, oozing/crusts, excoriations,lichenification and dryness, whereby dryness is evaluated on uninvolved areas;
  C: the subjective symptoms of pruritus at application areas and sleep loss evaluated on a visual analogue scale from 0 to 10 (average for the last three days or nights) and added. The intensity of each of the criteria erythema, edema/papulation, oozing/crusts, excoriations, lichenification and dryness will be graded according to the following 4 point scale:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe Each single parameter for SCORAD calculation will be documented on a source document. The SCORAD will be calculated according to the formula A/5 + 7B/2 + C and documented in the source documents and the CRF.

SECONDARY OUTCOMES:
The change from baseline in modified local SCORAD | On Days 3, 5, 8, and 12
Modified local SCORAD | on Days 1, 3, 5, 8, 12, and 15
  The intensity of each of the criteria will be graded according to the following 4 point scale and documented in the CRF:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe
Change from baseline in transepidermal water loss (TEWL) | On Days 3, 5, 8, 12, and 15
TEWL on Days 1, 3, 5, 8, 12, and 15 | Days 1, 3, 5, 8, 12, and 15
Subjective assessment of pruritus using a 10-point rating scale | Days 1, 3, 5, 8, 12, and 15
  Subjective assessment of pruritus at test sites on Days 1, 3, 5, 8, 12, and 15 using a 10-point rating scale.
Subjective efficacy assessment on Days 3, 5, 8, 12 and 15 | Days 3, 5, 8, 12 and 15
  The efficacy of the IMPs will be assessed in each test area by asking the patients using the following 5-point rating scale: The answer of the patients will be documented in the CRF.
  0 = no activity
  1. = poor
  2. = fair
  3. = good
  4. = excellent
Subjective dermal tolerability assessment using a 5-point rating scale on Days 3, 5, 8, 12 and 15 | Days 3, 5, 8, 12 and 15
  The dermal tolerability of the IMPs will be assessed in each test area by asking the patients using the following 5-point rating scale: The answer of the patients will be documented in the CRF.
  0 = no activity
  1. = poor
  2. = fair
  3. = good
  4. = excellent
Pharmacokinetic outcome measure | Day 1 and Day 15
  The pharmacokinetic endpoints are the hgd40 levels on Days 1 (pre-dose and 1, 2, 4 and 6 h post-dose) and 15 (pre-dose and 1, 2, 4 and 6 h post-dose and 24 h post-dose to Day 15).
Physical examination of the skin and Vital signs | Screening period and day 16
Adverse Events | Including the whole screening period and the experimental phase day -14 to day 16
Standard Safety laboratory | Screening period + on days 1, 5 and 16 in the Treatment period
  Including serology, IgE [immunoglobulin E] and sx1 test at screening

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Werfel, Prof. Dr., Principal Investigator — Division for Immunodermatology and Allergy Research Clinic for Dermatology, Allergy and Venereology Hannover Medical School
Locations (1):
- Division for Immunodermatology and Allergy Research Clinic for Dermatology, Allergy and Venereology Hannover Medical School, Hanover, Germany